CLINICAL TRIAL: NCT03243097
Title: Contralateral Routing of Signal in Unilateral Cochlear Implant Users
Brief Title: CROS Application in CI
Acronym: CROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hillary A Snapp, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20170029
Record Dates: First submitted 2017-06-07; First posted 2017-08-08 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Subjects (Experimental): All subjects enrolled in the study are required to complete Phase I before entering Phase II, and Phase II before entering Phase III.
  Interventions: Device: Phase I - Standard Microphone Cros Input; Device: Phase II - Automatic directional microphone Cros Input; Device: Phase III - No Cros Input

INTERVENTIONS:
Device: Phase I - Standard Microphone Cros Input — Subject will be fit with the research processor plus CROS microphone and wear for a 4 week period
Device: Phase II - Automatic directional microphone Cros Input — Automatic directional microphone technology will be activated in the research processor. Subjects will wear the CI+CROS configuration with directionality activated exclusively for 4-weeks.
Device: Phase III - No Cros Input — Subjects will return the research processor and CROS device and wear their own processor for a 2-week period

SUMMARY:
Bilateral profound sensorineural hearing loss (PSNHL) is often treated with Cochlear Implants. The majority of bilaterally deafened patients, however, often only receive a unilateral cochlear implant (CI), with resultant limitations related to monaural listening. For unilateral CI users, the deficits inherently associated with monaural listening remain despite the considerable benefits achieved through implantation. Providing bilateral input to monaural listeners (MLs) overcomes some of these disadvantages. Treatment by contralateral routing of signal (CROS) hearing aids, where the signal of interest is routed from the impaired (deaf) ear to the normal cochlea for processing is a promising alternative in unilateral CI recipients who cannot benefit from bilateral CIs. Utilizing CROS technology provides a less invasive alternative for patients who are unable or unwilling to undergo a second CI surgery and offers an innovative approach to resolving the auditory deficits associated with monaural listening. CROS technology has been used to treat traditional monaural listeners since 1965. When applied to unilateral CI users, this novel approach can overcome a key limitation of current treatment by restoring access to sound from the non-implanted ear and improving speech perception in noise.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Advanced Bionics CI recipient
* ≥ 6 months CI-listening experience and/or better than 50%-word recognition on Consonant-Nucleus-Consonant (CNC) word testing
* English speaking

Exclusion Criteria:

* Subjects who do not meet one or more of the above mentioned inclusion criteria are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Speech perception in noise | 8 weeks
  Speech perception in noise will be evaluated with the subjects cochlear implant alone and then with the combined application of CROS technology to the cochlear implant.

SECONDARY OUTCOMES:
Subjective Benefit | 8 weeks
  Benefit of wireless CROS technology with the cochlear implant will be assessed using a customized questionnaire with the subjects cochlear implant alone and then with the combined application of CROS technology to the cochlear implant.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Snapp, AuD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Department of Otolaryngology, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No